CLINICAL TRIAL: NCT06204016
Title: Associations of Estradiol and Stress Reactivity in Pre- and Postmenopausal Women
Brief Title: Estradiol and Stress Reactivity in Women
Status: Recruiting | Type: Observational
Sponsor: International Research Training Group 2804 (Other)
Collaborators: University Hospital Tuebingen (Other); German Research Foundation (Other); Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: IRTG_P02
Record Dates: First submitted 2023-12-21; First posted 2024-01-12 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Stress vs. Control; Estradiol vs. Placebo
Keywords: stress reactivity; mood homeostasis; neuroimaging (fMRI); menopause; menstrual cycle; sex hormones; women's mental health; estradiol
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- premenopausal women: naturally cycling women without hormonal contraception
  Interventions: Drug: Estradiol Valerate; Drug: Placebo
- postmenopausal women: women after menopause (min. 12 months no menstrual bleeding)
  Interventions: Drug: Estradiol Valerate; Drug: Placebo

INTERVENTIONS:
Drug: Estradiol Valerate — To elevate estradiol levels each woman will receive 12mg on two consecutive days (total 24mg) of estradiol valerate (Progynova21©)
  Other Names: Progynova21
Drug: Placebo — Placebo tablets will be administered as placebo-controlled condition (P-Tabletten White 7mm, Lichtenstein)
  Other Names: P-Tabletten

SUMMARY:
Stress reactivity and prevalence of stress related diseases differ between pre- and postmenopausal women. Thus, hormonal fluctuations may present a general vulnerability factor for stress-related diseases. Especially, the gonadal hormone estradiol (E2) seems to modulate the activity of stress related brain areas. The hippocampus and prefrontal areas control the amygdala's response to stress, and E2 may directly modulate the activity, connectivity and structure of these areas. In premenopausal women E2 seems to reduce stress reactivity. However, in postmenopausal women, who no longer produce E2 from the ovaries, E2 seem to increase stress reactivity. With the proposed study the investigators want to directly test E2's modulating effects (disentangled from other gonadal hormones) on stress reactivity of premenopausal women during their early follicular phase, and postmenopausal women by subjecting both groups of women to a psychosocial stress task in a neuroimaging environment.

DETAILED DESCRIPTION:
In a double-blinded repeated-measures within-between placebo-controlled design, two groups of women (premenopausal / postmenopausal) will receive either a placebo or estradiol valerate to experimentally increase estradiol (E2) levels. They will further undergo a psychosocial stress task (Montreal Imaging Stress Task) in a neuroimaging environment (functional magnetic resonance imaging - fMRI). By applying a multilevel approach, the investigators will be able to look at stress reactivity from a subjective, sympathetic (heart rate, skin conductance), endocrine (cortisol) and neural perspective. The investigators will further assess how changes in stress reactivity due to E2 increase are associated with gonadal hormones, and changes in neural activity, anatomy and connectivity in pre- compared to postmenopausal women.

At an initial screening session (T0) the investigators will be assessing sociodemographic variables, hand dominance, verbal intelligence, trial making, personality traits, gender identity and roles, childhood trauma, coping styles, sleep, female sexual health, reproductive status, menopausal symptoms, eating behaviour and premenstrual symptoms. After this all women will be invited to the first experimental session (T1, day 1), where blood and hair cortisol samples will be taken, subjective mood will be measured and the first pill treatment administered (placebo or E2 valerate, double-blinded) approx. 24h before the stress induction. They receive a second pill that they should take-in during the next day (T1/day2) approx. 4h before the stress induction. On T1/day 2 in the afternoon, participants come to the laboratory where the experimental procedure takes place. Participants will again be screened for MRI-exclusion criteria and after ensuring that all requirements are met to go into the MR-scanner, participants will be prepared (application of sensor for pulsoxymetry and electrodes for skin conductance assessment) and moved into the scanner, where they will undergo the stress induction via the Montreal Imaging Stress Task (MIST), a resting state scan, an anatomical scan and a diffusion tensor imaging (DTI) measurement. Throughout the MR-session, pulsoxymetry and skin conductance will constantly be assessed. Mood, subjective affect and stress, and saliva samples for further cortisol analyses will be taken at six time points throughout the experimental session. Furthermore, subjective variables on stress, self-esteem, emotion regulation, positive and negative affect, emotional self-rating, resting state, mental health, depression and anxiety scores and side effects of E2 intake will be assessed. A blood sample will be drawn (30ml) by medically trained personnel during the experimental session. For seven days following the experimental session, participants will give daily information on subjective experiences via an ecological momentary assessment (EMA). Then, the second experimental session (T2) will be scheduled at least two menstrual cycles (naturally cycling women) or 2 months (postmenopausal women) after the first experimental session (T1). For naturally cycling women, both experimental sessions will be scheduled up to 5 days after onset of menses. Naturally cycling women are asked to report the onset of their next menses after the experimental session. The procedure of the second experimental session (T2) will be similar to that of T1.

ELIGIBILITY:
Inclusion Criteria:

* Women, biologically female (assigned sex at birth)
* normal body mass index (18-28 kg/m2)
* Caucasian
* non-smoking
* German language fluency: at least advanced technical college entrance qualification
* Naturally cycling women, older than 18 years with a regular menstrual cycle (25-35 days) and postmenopausal women up to the age of 60 will be included.

Exclusion Criteria:

* Neurological or mental disease
* Medical problems such as hormonal, metabolic, or chronic diseases (e.g., severe hypertension, diabetes, dysfunctions of the thyroid, or congestive heart failure) as well as venous thromboembolism
* Pregnancy, delivery, and lactation (current and within the last year)
* Any kind of steroid hormonal, pharmacological treatment, or psychotropic treatment in the last three months
* Shift work
* Participants engaging in competitive/extreme sports
* Contraindication for MRI

  * People with non-removable metal objects on or in the body
  * Tattoos (if not MRI-incompatible according to expert guidelines)
  * Pathological hearing or increased sensitivity to loud noises
  * Claustrophobia
  * Surgery less than three months ago
  * Neurological disease or injury
  * Moderate or severe head injury
  * Intake of antidepressants or neuroleptics
  * Restricted vision

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will mainly consist of residents of Tübingen and surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Associations between elevated E2 concentration and acute stress effects on subjective experience | Measured twice two-three months apart; each time: approx. 45 minutes before stress onset, just before stress onset, immediately after stress, approx. 40 minutes, 60 minutes and 120 minutes after stress onset
  Ratings of positive and negative affect as well as stress, before and after stress induction. Comparing E2 against placebo in pre- and postmenopausal women.
Associations of E2 and acute stress effects on Hypothalamic-Pituitary-Adrenal-axis (HPA) response | Measured twice two-three months apart; each time: approx. 45 minutes before stress onset, just before stress onset, immediately after stress, approx. 40 minutes, 60 minutes and 120 minutes after stress onset
  Cortisol saliva samples before and after the stress task as indicator of stress/HPA-axis activation. Comparing E2 against placebo in pre- and postmenopausal women.
Association between E2 concentration and acute stress induced effects on neural level. | Measured twice three months apart; each time: approx. 5 minutes during neuroimaging
  Variability in activity of the brains stress network will be quantified using fMRI to assess differences between stress vs. control conditions during the stress task. Changes in activity will be assessed within regions associated with stress reactivity and regulation (amygdala, hippocampus, prefrontal cortex, anterior cingulate cortex (ACC), middle frontal gyrus (MFG), right superior temporal gyrus (STG), insula, striatum and praecuneus). Comparing E2 against placebo in pre- and postmenopausal women.
Association between E2 concentration and brain volume changes | Measured twice two- three months apart; each time: approx. 10 minutes during neuroimaging
  Via structural MRI scans changes in brain volume following E2 administration compared to placebo will be assessed, especially for the following brain regions: amygdala, hippocampus, prefrontal cortex (including orbito frontal cortex), anterior cingulate cortex (ACC), insula, middle frontal gyrus (MFG), right superior temporal gyrus (STG), fusiform gyrus, thalamus, cerebellum and inferior parietal lobule (IPL). Comparing E2 against placebo in pre- and postmenopausal women.
Association between E2 concentration and connectivity (resting state) changes | Measured twice two-three months apart; each time: approx. 10 minutes during neuroimaging
  Via a resting state scan, effects of estradiol concentration compared to placebo administration on connectivity changes will be assessed by applying whole brain network (especially Default Mode, Dorsal Attention, Frontoparietal, and Limbic networks) and region of interest analysis (especially of the amygdala, middle temporal gyrus (MTG), inferior frontal gyrus (IFG), postcentral gyrus, striatum, insula and ventrolateral, dorsolateral and medial prefrontal cortex (PFC), fusiform gyrus and anterior cingulate gyrus (ACC)). Comparing E2 against placebo in pre- and postmenopausal women.
Changes in hormonal levels induced by increased E2 concentration. | Measured twice two-three months apart; pill intake a day before and on the day of neuroimaging
  Changes in E2 levels (pmol/L) will be assessed from blood samples before and after pill intake (placebo or estradiol valerate) and stress induction. Comparing E2 against placebo in pre- and postmenopausal women.
Changes in hormonal levels induced by increased E2 concentration. | Measured twice two-three months apart; pill intake a day before and on the day of neuroimaging
  Changes in progesterone, testosterone, and allopregnanolone levels (nmol/L) will be assessed from blood samples before and after pill intake (placebo or estradiol valerate) and stress induction. Comparing E2 against placebo in pre- and postmenopausal women.

SECONDARY OUTCOMES:
Associations between E2 concentration and acute stress effects on physiological responses. | Measured twice two-three months apart; each time: 20 minutes during the fMRI stress task
  Measurements of heart rate and skin conductance as indicators of stress during fMRI. Comparing E2 against placebo in pre- and postmenopausal women. Comparing placebo against estradiol as well as pre- and postmenopausal women.
Association between E2 concentration and chronic stress | Measured twice two-three months apart
  Associations of chronic stress, assessed via hair cortisol measures and chronic stress questionnaire (Trier Inventar of Chronic Stress - TICS; value range = [0 228]; higher outcome relates to a higher chronic stress rating), with estradiol and stress reactivity. Comparing E2 against placebo in pre- and postmenopausal women.
Association between E2 concentration and effects on aftermath of stress. | Measured twice two-three months apart; each time for 7days
  To assess the subjective experience during the period following stress induction,an ecological momentary assessement EMA (7 days) will be obtained. Comparing E2 against placebo in pre- and postmenopausal women.
Associations between elevated E2 concentration and acute stress effects on subjective experience | Measured twice two-three months apart; each time: approx. 45 minutes before stress onset and120 minutes after stress onset
  Ratings of self-esteem before and after stress induction. Comparing E2 against placebo in pre- and postmenopausal women.
Associations between elevated E2 concentration and acute stress effects on subjective experience | Measured twice two-three months apart; each time: approx. 45 minutes before stress onset and120 minutes after stress onset
  Ratings of state anxiety before and after stress induction. Comparing E2 against placebo in pre- and postmenopausal women.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Derntl, Prof., Principal Investigator — Departement of Psychiatry & Psychotherapy
Locations (1):
- University of Tuebingen; Department of Psychiatry & Psychotherapy, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
After publication and finishing the study, anonymized research data cab be available.
Time Frame: Data can become available after an embargo period of 12 months after completion and publication of the study
Access Criteria: Researchers may contact the lead PI to gain access